CLINICAL TRIAL: NCT06150963
Title: Virtual Reality for the Management of Pain and Anxiety for Outpatient Interventional Radiology Procedures Performed With Local Anesthesia: A Randomized Pilot Study in Digital Sedation
Brief Title: Virtual Reality for the Management of Pain and Anxiety for Outpatient Interventional Radiology Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 27238
Record Dates: First submitted 2023-11-12; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pain; Anxiety
Keywords: Interventional Radiology; Thyroid Biopsy; Peripherally Inserted Central Catheter; Virtual Reality; Pain; Anxiety; Visual Analog Scale
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Thyroid Biopsy (Control) (Active Comparator): Patients within this arm received standard procedure thyroid biopsies without virtual reality.
  Interventions: Procedure: Standard Procedure Thyroid Biopsy
- Thyroid Biopsy (Virtual Reality) (Experimental): Patients within this arm received standard procedure thyroid biopsies with virtual reality for the length of the procedure.
  Interventions: Device: Virtual Reality; Procedure: Standard Procedure Thyroid Biopsy
- PICC (Control) (Active Comparator): Patients within this arm received standard procedure PICC placements without virtual reality.
  Interventions: Procedure: Standard Procedure PICC Placement
- PICC (Virtual Reality) (Experimental): Patients within this arm received standard procedure PICC placements with virtual reality for the length of the procedure.
  Interventions: Device: Virtual Reality; Procedure: Standard Procedure PICC Placement

INTERVENTIONS:
Device: Virtual Reality — Study participants assigned to the VR intervention group were fitted with an HP Reverb G2 Head Mounted Display (HMD) and a wireless mouse prior to preparation for procedure. One virtual environment was utilized, integrating passive and active participant input via gyroscopic motion detection and computer mouse input.
  Arms: PICC (Virtual Reality); Thyroid Biopsy (Virtual Reality)
Procedure: Standard Procedure Thyroid Biopsy — In this procedure the patient lies down on a bed with their neck tilted back to reveal the thyroid gland. The doctor cleans the skin over the nodule and numbs it with a local anesthetic. The doctor will then use an ultrasound device to visualize the nodule and guide a needle to obtain cells through the syringe. This process may be repeated several times to retrieve adequate tissue for analysis.
  Arms: Thyroid Biopsy (Control); Thyroid Biopsy (Virtual Reality)
Procedure: Standard Procedure PICC Placement — In this procedure the patient lies down on a bed and has their arm cleaned and then numbed with a local anesthetic. The doctor then uses an ultrasound to locate a suitable vein in the arm, typically above the elbow. The physician then makes a small incision in the skin and inserts a needle into the vein, followed by guidance of the Peripherally Inserted Central Catheter (PICC) through the needle until it reaches a large vein near the heart. The final position is confirmed by X-ray and the PICC line is secured at the site of insertion.
  Arms: PICC (Control); PICC (Virtual Reality)

SUMMARY:
This study explores the use of virtual reality (VR) to reduce pain and anxiety during thyroid biopsies and PICC line insertions under local anesthesia. One group experienced the procedure with VR, while the other group did not. Participants completed questionnaires before and after the surgery to measure pain and anxiety levels. The main goal is to observe if VR can significantly decrease pain and anxiety during these procedures.

DETAILED DESCRIPTION:
This prospective, randomized, controlled study investigates the efficacy of virtual reality (VR) as a means to alleviate pain and anxiety in individuals receiving thyroid biopsies and PICC placements with local anesthesia. This study was conducted at Temple University Hospital between June 2021 and August 2022. A total of 107 patients were randomized into treatment and control groups. The VR experience involved wearing a headset with an immersive 3D visual display and accompanying music, simulating a calming environment. Patients completed Visual Analog Scales for pain and anxiety both before and after the intervention, reflecting their pain and anxiety levels prior to and during the procedure. The primary endpoints were to observe the effect of VR on pain and anxiety in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Scheduled to receive Fine-Needle Aspiration (FNA) Thyroid Biopsy
* Scheduled to receive Peripherally Inserted Central Catheters (PICC)

Exclusion Criteria:

* Declining to participate
* Inability to provide consent
* Emergency procedures
* Administration of general anesthesia/moderate sedation
* Visual or hearing deficits
* Pregnancy
* Current prisoner status
* Nerve or sensory deficits over area of procedure
* COVID-19 positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | Immediately prior to and after procedure
  Pre-procedure pain assessments were obtained using a Visual Analog Scale (VAS) corresponding to the patient's expected level of pain during each procedure prior to randomization to treatment or control. VAS scale was measured in mm, 0mm indicating "no pain", 100mm indicating "worst pain." Following each procedure, participants completed a self-reported survey indicating actual pain felt during procedure on VAS scale.
Anxiety (VAS) | Immediately prior to and after procedure
  Pre-procedure anxiety assessments were administered using a VAS scale to indicate the patient's level of anxiety prior to randomization to treatment or control. Similar to pain, VAS anxiety scale was measured in mm, 0mm indicating "no anxiety", 100mm indicating "worst anxiety." Following each procedure, participants completed a self-reported survey indicating actual level anxiety experienced during the procedure on VAS scale.

SECONDARY OUTCOMES:
Pulse Rate (bpm) | Three times during procedure
  Pulse rate was monitored and collected at three points during each trial: immediately after headset placement, six minutes into the procedure, and immediately following completion of the procedure.
Systolic Blood Pressure (mmHg) | Three times during procedure
  Systolic blood pressure was collected at three points during each trial: immediately after headset placement, six minutes into each procedure, and immediately following completion of the procedure.
Diastolic Blood Pressure (mmHg) | Three times during procedure
  Diastolic blood pressure was collected at three points during each trial: immediately after headset placement, six minutes into each procedure, and immediately following completion of the procedure.
Procedure Length | Duration of procedure
  Procedure length recorded in minutes
Lidocaine Administered | Immediately after procedure
  Quantity of subcutaneous lidocaine administered recorded in milliliters (mL).

CONTACTS AND LOCATIONS:
Overall Officials: Hillel Maresky, M.D., Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results reported in the main publication, including demographics, outcomes, and adverse events, will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 5 years.
Access Criteria: Access to trial IPD can be requested by qualified research engaging in independent scientific research, and will be provided following review and approval of a research proposal and a data sharing agreement.

REFERENCES:
- [Result] Mallari B, Spaeth EK, Goh H, Boyd BS. Virtual reality as an analgesic for acute and chronic pain in adults: a systematic review and meta-analysis. J Pain Res. 2019 Jul 3;12:2053-2085. doi: 10.2147/JPR.S200498. eCollection 2019. PMID 31308733
- [Result] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481